CLINICAL TRIAL: NCT04946448
Title: COmbinAtion Therapy of dieT With biologicalS for Crohn's Disease: the OATS Study
Acronym: OATS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S64746
Record Dates: First submitted 2021-06-18; First posted 2021-06-30 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Crohn Disease; Inflammatory Bowel Diseases; Diet, Healthy
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FIT group (Experimental): Patients treated with biological treatment and the FIT diet
  Interventions: Other: FIT diet
- Control group (No Intervention): Patients treated with biological treatment and the standard diet

INTERVENTIONS:
Other: FIT diet — Dietary intervention as add-on therapy to biologicals
  Arms: FIT group

SUMMARY:
This study is a randomised open label study, comparing the FIT diet with standard diet in patients with Crohn's disease treated with biologic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18-80 years)
* active inflammation of terminal ileum and/or colon with a Simple Endoscopic Score for Crohn's Disease (SES-CD) greater than 5 (or greater than 3 for patients with isolated ileitis),
* patient reported outcome 2 (PRO2 - 7 day average daily stool frequency x 2 + 7 day average daily abdominal pain score x 5) > 8,
* faecal calprotectin above 250 µg/g.

Exclusion Criteria:

* Abcess,
* Bowel resection within 6 months before enrolment,
* Ostomy,
* Short-bowel syndrome,
* Clinically significant stricture that could require surgery,
* Pregnant,
* Lactating woman or desire to become pregnant during the study,
* Unwilling or unable to follow the study diet.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2021-09-14 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Steroid-free clinical and biochemical remission | Month 6
  Normalization of faecal calprotectin (< 250 µg/g) and steroid-free clinical remission, defined as patient PRO2 ≤ 8 (average daily stool frequency ≤ 1.5 AND average daily abdominal pain score ≤ 1), at month 6.

SECONDARY OUTCOMES:
Clinical response | 6 months and 1 year
  ≥ 30% decrease in average daily stool frequency and/or ≥ 30% decrease in average daily abdominal pain score and both not worse than baseline
Clinical remission | 6 months and 1 year
  PRO2≤8
Steroid-free clinical remission | 6 months and 1 year
  PRO2≤8, no steroids
Endoscopic remission | 1 year
  SES-CD <2
Endoscopic improvement | 1 year
  drop in SES-CD with at least 50%
CRP improvement | 6 months and 1 year
  50% or more improvement in CRP or CRP <5 mg/L
Fecal calprotectin improvement | 6 months and 1 year
  50% or more improvement in faecal calprotectin or faecal calprotectin <250 µg/g
Number of participants without nutritional deficiencies | 6 months and 1 year
  Absence of vitamin B12, vitamin D, folic acid, iron deficiencies
Fatigue | 6 months and 1 year
  30% or more improvement in IBD Disk energy score
Health-related quality of life | 6 months and 1 year
  30% or more improvement in overall IBD Disk score

CONTACTS AND LOCATIONS:
Overall Officials: João PG Sabino, MD PhD, Principal Investigator — UZ Leuven
Locations (1):
- University Hospital of Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No